CLINICAL TRIAL: NCT00365755
Title: Comparison of High Dose Rapid Schedule With Conventional Schedule Chemotherapy for Stage 4 Neuroblastoma Over the Age of One Year
Brief Title: Combination Chemotherapy in Treating Young Patients Who Are Undergoing Surgery and an Autologous Bone Marrow Transplant for Disseminated Neuroblastoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CCLG-ENSG-5; CDR0000454576 (Registry Identifier: PDQ (Physician Data Query)); EU-20592; CCLG-NB-1990-11
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2008-03

CONDITIONS: Neuroblastoma
Keywords: disseminated neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Carboplatin; Cisplatin; Cyclophosphamide; Etoposide; Melphalan; Vincristine

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Drug: cyclophosphamide
Drug: etoposide
Drug: melphalan
Drug: vincristine sulfate
Procedure: autologous bone marrow transplantation
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Giving combination chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. A bone marrow transplant, using bone marrow from the patient, may be able to replace blood-forming cells that were destroyed by chemotherapy. It is not yet know which combination chemotherapy schedule is more effective, when given before surgery and an autologous bone marrow transplant, in treating patients with disseminated neuroblastoma.

PURPOSE: This randomized phase III trial is studying two different chemotherapy schedules to compare how well they work in treating young patients who are undergoing surgery and an autologous bone marrow transplant for disseminated neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the response rates (bone marrow and primary tumor) in young patients with disseminated neuroblastoma treated with two different combination chemotherapy schedules comprising vincristine, cyclophosphamide, cisplatin, etoposide, and carboplatin followed by surgery and autologous stem cell transplantation.
* Compare the event-free survival of patients treated with these regimens.
* Compare the prognostic factors of patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I (OPEC/OJEC): Patients receive OPEC combination chemotherapy comprising vincristine IV, cyclophosphamide IV, cisplatin IV continuously over 24 hours, and etoposide IV over 4 hours on day 1 of course 1. Patients then receive OJEC combination chemotherapy comprising vincristine IV, cyclophosphamide IV, etoposide IV over 4 hours, and carboplatin IV over 1 hour on day 1 of course 2. OPEC and OJEC regimens alternate so that patients receive 4 courses of OPEC and 3 courses of OJEC over 18 weeks in the absence of disease progression or unacceptable toxicity.
* Arm II (Rapid COJEC): Patients receive vincristine IV and carboplatin IV over 1 hour on day 1 and etoposide IV over 4 hours on days 1 and 2 (regimen 1). Ten days later, patients receive vincristine IV followed by cisplatin IV continuously over 24 hours on day 1 (regimen 2). Ten days later, patients receive vincristine IV on day 1 and etoposide IV over 4 hours and cyclophosphamide IV on days 1 and 2 (regimen 3). Treatment continues for 10 weeks (with a 10-day interval between regimens in this order: regimen 2, regimen 1, regimen 2, regimen 3, and regimen 2) in the absence of disease progression or unacceptable toxicity.

Patients who achieve bone marrow complete remission then undergo surgery. Patients achieving bone marrow partial remission or less are removed from study.

After surgery, patients receive cyclophosphamide IV on day -7 and undergo bone marrow harvest on day 1. Patients then receive high-dose melphalan IV on day 1. Autologous bone marrow cells are reinfused on day 3.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 190 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed disseminated neuroblastoma

  * No local or regional neuroblastoma
  * No disseminated disease that is demonstrated by meta-iodobenzylguanidine (MIBG) scan only
* Needle biopsy of primary tumor required

  * Fine needle aspiration is not adequate

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy
* No other prior therapy

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Ross Pinkerton, MD — Royal Marsden NHS Foundation Trust; Andrew David J. Pearson, MD, FRCP, DCh, Study Chair — University of Newcastle Upon-Tyne; Ian J. Lewis, MD — Leeds Cancer Centre at St. James's University Hospital

REFERENCES:
- [Result] Pearson AD, Pinkerton CR, Lewis IJ, Imeson J, Ellershaw C, Machin D; European Neuroblastoma Study Group; Children's Cancer and Leukaemia Group (CCLG formerly United Kingdom Children's Cancer Study Group). High-dose rapid and standard induction chemotherapy for patients aged over 1 year with stage 4 neuroblastoma: a randomised trial. Lancet Oncol. 2008 Mar;9(3):247-56. doi: 10.1016/S1470-2045(08)70069-X. PMID 18308250
- [Derived] Moreno L, Vaidya SJ, Pinkerton CR, Lewis IJ, Imeson J, Machin D, Pearson AD; European Neuroblastoma Study Group; Children's Cancer and Leukaemia Group (CCLG) (formerly UKCCSG). Long-term follow-up of children with high-risk neuroblastoma: the ENSG5 trial experience. Pediatr Blood Cancer. 2013 Jul;60(7):1135-40. doi: 10.1002/pbc.24452. Epub 2012 Dec 31. PMID 23281263